CLINICAL TRIAL: NCT04700618
Title: A Phase Ⅳ Clinical Trial to Evaluate the Safety and Immunogenicity of 23 Valent Pneumococcal Polysaccharide Vaccine Revaccinated in 60-70 Years Old in Shanghai
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of PPV23 Vaccine Revaccinated in 60-70 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Shanghai Municipal Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PPV23-2021-2
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Vaccination
Keywords: safety; immunogenicity
MeSH Terms: interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Intervention Model Description: Study group is PPV23 revaccination and control group PPV23-vaccination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The subjects in the study group had been vaccinated with 23 valent pneumococcal polysaccharide vaccine made in China for more than 5 years.
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine
- Control group (Placebo Comparator): The control group had never been vaccinated with any pneumococcal vaccine.
  Interventions: Biological: 23-valent pneumococcal polysaccharide vaccine

INTERVENTIONS:
Biological: 23-valent pneumococcal polysaccharide vaccine — The study group and the control group were vaccinated with one dose of vaccine and blood was collected after 28-40 days.

SUMMARY:
Objective: To evaluate the safety and immunogenicity of PPV23 vaccine revaccinated in 60-70 years old in Shanghai.

DETAILED DESCRIPTION:
1. Antibody double growth rate in 28-40 days after immunization;
2. Antibody GMC level in 28-40days after immunization;
3. Incidence of adverse reactions in 0-30days.

ELIGIBILITY:
Inclusion Criteria:

1. The age was 60-70 years old on the day of enrollment;
2. The subjects have signed the informed consent and signed the date;
3. The subjects are able to participate in all planned follow-up visits and were able to follow all trial procedures (e.g. complete diary card / contact card, return to visit);
4. The subjects in the study group had been vaccinated with 23 valent pneumococcal polysaccharide vaccine made in China for more than 5 years;
5. The control group had never been vaccinated with any pneumococcal vaccine; 6.Axillary temperature ≤37.0℃.

Exclusion Criteria:

1. With a medical history with hypersensitiveness, eclampsia, epilepsy, cerebropathia and neurological illness;
2. Allergic to any ingredient of vaccine or with allergy history to any vaccine; 3.Subjects with immunodeficency or suspected impairment of immunologic function (e.g. caused by HIV), or subjects are in the process of immunosuppressor therapy(Taking orally injecting of steroid hormone);

4.Administration of immunoglobulins within 30 days prior to this study; 5.Acute febrile disease(temperature ≥ 37.0°C) or infectious disease; 6.With a clearly diagnosed history of thrombocytopenia or other coagulopathy, may cause contraindications for subcutaneous injection; 7.With any serious chronic illness, acute infectious diseases, or respiratory diseases; 8.Suffering from serious cardiovascular diseases (pulmonary heart disease, pulmonary edema, hypertension can not be controlled to normal by drugs), liver and kidney diseases, diabetes with complications; 9.With any kind of infectious, purulent, or allergic skin diseases; 10.With any other factor that makes the investigator determines the subject is unsuitable for this study.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2022-02-13 (Actual)

PRIMARY OUTCOMES:
Antibody doubling rate | The blood collection time was 28-40 days after vaccination.
  The difference of serum antibody double growth level between the two groups was compared.

SECONDARY OUTCOMES:
Antibody GMC level | The blood collection time was 28-40 days after vaccination.
  The difference of serum antibody GMC level between the two groups was compared.
Incidence of adverse reactions | Within 30 days after vaccination.
  Adverse reactions were collected during the observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Guo, Study Chair — Shanghai Municipal Center for Disease Control and Prevention
Locations (1):
- Shanghai municipal center for disease control and prevention, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No